CLINICAL TRIAL: NCT03164694
Title: A Multicenter Phase II Trial of Pemetrexed Plus Carboplatin With or Without Apatinib in Patients With Advanced Non-small Cell Lung Cancer Without EGFR Mutation, ALK Gene Rearrangement, and ROS1 Gene Rearrangement
Brief Title: APatinib Plus Chemotherapy vErsus Chemotherapy As First-line Treatment for Advanced NSCLC
Acronym: APPEAL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1006
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — apatinib; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib (Experimental): Patients were given pemetrexed (500 mg/m2) plus carboplatin (AUC =5) plus apatinib. Apatinib was given 850 mg per day orally at day one of chemotherapy.
  Interventions: Drug: Apatinib; Drug: Pemetrexed; Drug: Carboplatin
- Control (Active Comparator): Patients were given pemetrexed (500 mg/m2) plus carboplatin (AUC =5).
  Interventions: Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Apatinib — Apatinib was given 850 mg per day orally.
  Arms: Apatinib
Drug: Pemetrexed — pemetrexed (500 mg/m2)
Drug: Carboplatin — carboplatin (AUC =5)

SUMMARY:
The purpose of this study is to studying the addition of apatinib with chemotherapy to investigate the efficacy and safety of apatinib in combination with chemotherapy in patients with advanced NSCLC.

DETAILED DESCRIPTION:
Platinum-based chemotherapy is the recommended therapeutic approach for patients with advanced non-small cell lung cancer (NSCLC) without EGFR mutation, ALK gene rearrangement, and ROS1 gene rearrangement. However, the prognosis of advanced NSCLC remains poor. Apatinib is a novel tyrosine kinase inhibitor targeting vascular endothelial growth factor receptor-2. Apatinib has been proved to be effective and safe in heavily pretreated patients with gastric cancer. This study is to studying the addition of apatinib with chemotherapy to investigate the efficacy and safety of apatinib in combination with chemotherapy in patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Target population is advanced NSCLC (IIIB-IV) without EGFR mutation, ALK gene rearrangement, and ROS1 gene rearrangement.
* Written informed consent provided.
* Male and female patients aged ≥18 years, < 75 years.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Life expectancy ≥12 weeks.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
* Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Known severe hypersensitivity to apatinib or any of the excipients of this product.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
* Patients with prior chemotherapy or therapy with systemic anti-tumour therapy (e.g. monoclonal antibody therapy).
* Patients with prior radiotherapy
* History of another malignancy in the last 5 years with the exception of the following: other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Eye inflammation or eye infection not fully treated or conditions predisposing the subject to this.
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.
* Patient who has active serious infection (e.g. pyrexia of or 38.0℃ over)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year after the last patient is randomized
  Overall survival was assessed from randomization to death as a result of any cause.

SECONDARY OUTCOMES:
Disease-free survival | 1 year after the last patient is randomized
  Disease-free survival was assessed from randomization to disease recurrence or death as a result of any cause.
Number of Participants with Adverse Events | 1 year
  To assess if the addition of apatinib to chemotherapy is safe.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China